CLINICAL TRIAL: NCT00837369
Title: Regadenoson Real Time Perfusion Imaging Trial
Brief Title: Regadenoson R-T Perfusion Imaging Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Mayo Clinic (Other); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0566-08-FB
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Myocardial Perfusion Abnormalities
Keywords: Stress echocardiography; SPECT; Myocardial perfusion imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson; perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 Real time perfusion (RTPE) imaging following Regadenoson (Experimental): RTPE studies (resting and following Regadenoson 400 ug IV bolus injection) will be performed during a continuous infusion of lipid encapsulated microbubbles (Definity, Lantheus Medical Imaging) to qualitatively and quantitatively examine wall motion and myocardial contrast enhancement.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — 400ug IV bolus injection, single dosage
  Other Names: Definity (Lantheus Medical Imaging); Lipid encapsulated microbubbles

SUMMARY:
To exam the feasibility and accuracy of Regadenoson real time perfusion (RTPE) Imaging during vasodilator stress with Regadenoson for detection of significant coronary artery disease (CAD) in patients scheduled to undergo coronary angiography.

DETAILED DESCRIPTION:
To exam the feasibility and accuracy of RTPE during vasodilator stress with 400micrograms of the adenosine receptor (A2A) agonist Regadenoson for detection of significant coronary artery disease (CAD) in patients scheduled to undergo coronary angiography. Sensitivity, specificity , and accuracy of perfusion and wall motion analysis to identify a coronary stenosis> 50% in diameter by quantitive angiography will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Age ≥30 years.
* Resting Left Ventricular Ejection Fraction > 40% using Simpson's biplane measurement.
* Scheduled for coronary angiography within 30 days of the Regadenoson stress test.
* Negative urine pregnancy test within 2 hours of ultrasound contrast administration required of females of childbearing age unless post-menopausal or with evidence of surgical sterilization.
* Be conscious and coherent, and able to communicate effectively with trial personnel.
* Agreeable to undergo the additional stress test and coronary angiography
* Have at least an intermediate likelihood of coronary disease based on the following clinical profile
* Good apical echo images with at least 50% of each coronary artery territory well visualized.

Exclusion Criteria:

* Known or suspected hypersensitivity to ultrasound contrast agent used for the study.
* Pregnancy or lactation.
* Complicated hemodynamic instability (i.e., New York Heart Association (NYHA) Class IV heart failure, unstable angina at rest despite medical therapy).
* Life expectancy of less than two months or terminally ill.
* Congestive (idiopathic) or hypertrophic cardiomyopathy.
* Known left main disease.
* Heart transplant recipient, hypertrophic cardiomyopathy, acute myo- or pericarditis.
* Resting Left Ventricular Ejection Fraction < 40%
* Large inducible perfusion defects or wall motion abnormalities during prior stress imaging study associated with left ventricular cavity dilatation.
* Early positive treadmill EKG within the first stage of the test.
* History of >1st degree heart block, sick sinus syndrome or high grade atrioventricular (AV) block without a pacemaker.
* Dipyridamole use within 30 hours of stress test, or consumption of methylxanthines within 12 hours, or use of sublingual nitroglycerin within two hours.
* Participation In another investigational study within one month of this study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04-07 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medicial Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Groups:
- Regadenoson 400 ug IV Bolus Injection: Real time perfusion (RTPE) studies (resting and following Regadenoson 400 ug IV bolus injection) will be performed during a continuous infusion of lipid encapsulated microbubbles (Definity, Lantheus Medical Imaging) to qualitatively and quantitatively examine wall motion and myocardial contrast enhancement.
  Regadenoson: 400ug IV bolus injection, single dosage
Period: Overall Study
Arm/Group | Regadenoson 400 ug IV Bolus Injection
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Regadenoson: RTPE studies (resting and following Regadenoson 400 ug IV bolus injection) will be performed during a continuous infusion of lipid encapsulated microbubbles (Definity, Lantheus Medical Imaging) to qualitatively and quantitatively examine wall motion and myocardial contrast enhancement.
  Regadenoson: 400ug IV bolus injection, single dosage
Arm/Group | Regadenoson
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Detection of Coronary Artery Disease With Real-time Perfusion Echocardiography During Regadenoson Stress
Description: Regadenoson real-time myocardial contrast echocardiography can be used to detect coronary artery stenosis during Regadenoson stress.
Time Frame: 1 hour observation post perfusion
Population: 60 Males, 40 Females being evaluated for coronary artery disease.
Measure: Count of Participants; unit: Participants
Groups:
- Wall Motion: RTPE studies (resting and following Regadenoson 400 ug IV bolus injection) will be performed during a continuous infusion of lipid encapsulated microbubbles (Definity, Lantheus Medical Imaging) to qualitatively and quantitatively examine wall motion.
  Wall motion was assessed by scoring as follows: 1=normal, 2=hypokinetic, 3=akinetic, and 4=dyskinetic.
  An inducible wall motion abnormality was one in which a new wall motion abnormality was evident after regadenoson bolus within at least 2 contiguous segments. A fixed defect was one in which the abnormality,was present at rest and did not change after the regadenoson bolus.
- Myocardial Perfusion: RTPE studies (resting and following Regadenoson 400 ug IV bolus injection) will be performed during a continuous infusion of lipid encapsulated microbubbles (Definity, Lantheus Medical Imaging) to qualitatively and quantitatively examine myocardial perfusion.
  Myocardial perfusion was assessed by examination of myocardial contrast replenishment after brief high mechanical index impulses. A perfusion defect was defined as a delay (>2 seconds) in myocardial contrast replenishment in 2 contiguous segments.
Arm/Group | Wall Motion | Myocardial Perfusion
Number analyzed (Participants) | 100 | 100
Participants | 98 | 98
Statistical Analysis 1: Comparison: Wall Motion vs Myocardial Perfusion; Test type: Superiority; p < 0.001, Chi-squared — Compare the differences in sensitivity between myocardial perfusion and wall motion for detecting stenosis
Statistical Analysis 2: Comparison: Wall Motion vs Myocardial Perfusion; Test type: Superiority; p < 0.001, Chi-squared — Compare the sensitivity of myocardial perfusion in detecting stenosis within the first 4 minutes after regadenoson bolus injection to that of wall motion

ADVERSE EVENTS:
Time Frame: 1 hour observation
Description: Non-serious adverse persisted no more than 5 minutes for chest pain, shortness of breath & back pain. Headaches were reported within 1 hour.
Groups:
- Arm One: RTPE studies (resting and following Regadenoson 400 ug IV bolus injection) will be performed during a continuous infusion of lipid encapsulated microbubbles (Definity, Lantheus Medical Imaging) to qualitatively and quantitatively examine wall motion and myocardial contrast enhancement.
  Regadenoson: 400ug IV bolus injection, single dosage
  Non-serious adverse effects during Regadenoson and Definity administration included chest pain in 7% of patients, shortness of breath in 48%, headache in 23% and back pain in 4%.
Arm/Group | Arm One
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 82/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm One (N=100)
Chest Pain (Cardiac disorders) | 7 (7) — Chest Pain
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 48 (48) — Shortness of Breath
Headache (Vascular disorders) | 23 (23) — Headache
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) — Back pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No